CLINICAL TRIAL: NCT06355752
Title: Changes in Biomarkers of Pain and Stress Perception After the Application of a Dry Needling Technique in Patients With Low Back Pain
Brief Title: Biomarkers of Pain and Stress Perception and Dry Needling Technique Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Principal investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 0018-N-23
Record Dates: First submitted 2024-04-04; First posted 2024-04-09 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Dry needling; Biochemical Markers
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real dry needling (Experimental): Subjects included in this group will receive a session with dry needling in the quadratus lumborum muscle.
  Interventions: Other: Dry needling of lumbar iliocostalis muscle
- Sham dry needling (Sham Comparator): Subjects included in this group will receive a session with sham dry needling in the quadratus lumborum muscle.
  Interventions: Other: Sham dry needling lumbar iliocostalis muscle

INTERVENTIONS:
Other: Dry needling of lumbar iliocostalis muscle — Subjects will be treated with dry needling to the quadratus lumborum muscle. To do this, the subject will be lying laterally on the contralateral side and with the hip in an adducted position. Ten incisions will be made in the muscle.
  The head will rest comfortably on a pillow
  Arms: Real dry needling
Other: Sham dry needling lumbar iliocostalis muscle — Subjects will be treated with dry needling to the quadratus lumborum muscle. To do this, the subject will be lying laterally on the contralateral side and with the hip in an adducted position. The placebo needle will move 10 times imitating the real procedure.
  The head will rest comfortably on a pillow
  Arms: Sham dry needling

SUMMARY:
The use of the dry needling technique has become widespread in recent years for the treatment of musculoskeletal pain. Although dry needling has been shown to be effective in the treatment of shoulder pain, elbow pain, headache, etc., we do not yet have a clear understanding of the mechanisms of action that justify its beneficial effects.

In this study, we propose to analyse the biochemical markers of pain generated by the application of a dry needling technique on the lumbar musculature in patients with mechanical lumbar pain of non-specific origin.

The aim of this study will be to evaluate the effects of dry needling technique on the plasmatic concentration of biochemical markers.Furthermore, the test subjects will be randomly distributed into two groups.

An experimental group where the subjects will receive a real dry needling technique.

Another group will be treated with a sham technique.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical lumbar pain of more than three months of evolution.

Exclusion Criteria:

* Medical diagnosis of lumbar disc herniation or protrusion.
* Low back and leg pain.
* Pregnancy.
* Fibromyalgia.
* Fear of needles.
* Medication with anticoagulants

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-04-12 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Extracting Blood Samples and Obtaining Serum/Plasma | Change from Baseline concentration at 2 hours
  Serum samples will be extracted by venipuncture at the cubital fossa, according to a standardized protocol. Blood will be collected in a tube for serum (Vacutainer SST II Advance, model 367953) and a tube for plasma (Vacutainer PST II Advance, model 367374) separation. Substances related to antinociception will be determined later: Dopamine, adrenaline, norepinephrine, cortisol.

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Gallego-Izquierdo, PhD, Study Chair — Centro de Investigación Fisioterapia y Dolor
Locations (1):
- Centro Investigación Fisioterapia y Dolor, Alcalá de Henares, Madrid, Spain